CLINICAL TRIAL: NCT00637130
Title: Safety and IOP Lowering Efficacy of Low Dose Travoprost Ophthalmic Solutions Dosed BID Compared to TRAVATAN® in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Intraocular Pressure (IOP) Lowering Efficacy of Low Dose Travoprost
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-06-11
Record Dates: First submitted 2008-02-29; First posted 2008-03-17 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Travoprost 0.0008% (Experimental): Travoprost ophthalmic solution, 0.0008%, one drop in study eye(s) twice daily (8 AM and 8 PM), for 2 weeks
  Interventions: Drug: Travoprost ophthalmic solution, 0.0008%
- Travoprost 0.001% (Experimental): Travoprost ophthalmic solution, 0.001%, one drop in study eye(s) twice daily (8 AM and 8 PM), for 2 weeks
  Interventions: Drug: Travoprost ophthalmic solution, 0.001%
- Travoprost 0.0012% (Experimental): Travoprost ophthalmic solution, 0.0012%, one drop in study eye(s) twice daily (8 AM and 8 PM), for 2 weeks
  Interventions: Drug: Travoprost ophthalmic solution, 0.0012%
- TRAVATAN + Vehicle (Active Comparator): TRAVATAN, one drop in study eye(s) once daily (8 PM), and Vehicle, one drop in study eye(s) once daily (8 AM), for two weeks
  Interventions: Drug: TRAVATAN; Other: Vehicle
- Vehicle (Placebo Comparator): Vehicle, one drop in study eye(s) twice daily (8 AM and 8 PM), for 2 weeks
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Travoprost ophthalmic solution, 0.0008%
  Arms: Travoprost 0.0008%
Drug: Travoprost ophthalmic solution, 0.001%
  Arms: Travoprost 0.001%
Drug: Travoprost ophthalmic solution, 0.0012%
  Arms: Travoprost 0.0012%
Drug: TRAVATAN
  Arms: TRAVATAN + Vehicle
Other: Vehicle
  Arms: TRAVATAN + Vehicle; Vehicle

SUMMARY:
The purpose of this study is to compare the safety and IOP-lowering efficacy of various low dose travoprost formulations in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older, either sex or race with open-angle glaucoma or confirmed ocular hypertension
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Age related
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure | Up to 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center at 1-888-451-3937, Fort Worth, Texas, United States